CLINICAL TRIAL: NCT05770297
Title: Effect of Propolis Administration as Levonorgestrel (LNG) Implant Adjuvant for Dysmenorrhea in Endometriosis: Focus on Clinical Improvement, Oxidative Stress Biomarkers and Inflammation
Brief Title: Effect of Propolis Administration for Dysmenorrhea in Endometriosis Patient With Levonorgestrel Implant Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dr. drg. Dwirini Retno Gunarti, M.S., Head of Biochemistry Laboratory, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KET-683/UN2.F1/ETIK/PPM.00.02
Record Dates: First submitted 2023-01-24; First posted 2023-03-15 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Endometriosis; Dysmenorrhea
Keywords: Levonorgestrel implant; Propolis; Oxidative stress
MeSH Terms: conditions — Endometriosis; Dysmenorrhea | interventions — Propolis; caramel coloring; Ethanol

STUDY DESIGN:
Intervention Model Description: Endometriosis patients with menstrual pain who received LNG implant therapy were divided into two groups, each group consisted of 12 samples. The control group only received LNG, the treatment group received LNG with the addition of propolis. Propolis is given 2 times a day, namely in the morning before breakfast and at night before going to bed, with a dose of 1 drop /10 kg body weight (kgBW). Both groups were followed and reassessed after 1 month, 3 months both clinical and laboratory. Prior to receiving therapy, all subjects received education and signed informed consent for their willingness to participate in the study
Who Masked: Participant, Investigator
Masking Description: there will be a comparison group that will receive intervention in the same amount, preparation, and form, but only contain a placebo in the form of a 70% caramel alcohol dye solution. Investigator and participant will not know the contain of intervention that has given.
  Randomization of participants was carried out based on the arrival of participants to the obstetrics and gynecology clinic at the Cipto Mangunkusumo Hospital by labeling A for the intervention group and B for the treatment group. then data collection is carried out according to research procedures
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Propolis (Active Comparator): the subjects were asked to consume propolis 1 drop/10 kgbw/time given 2 times a day for 12 weeks. the dose will be calculated based on body weight by the certified nutritionist during the interview after the subject signs the informed consent form
  Interventions: Dietary Supplement: Propolis
- Placebo (Placebo Comparator): the subjects were asked to consume placebo (glucose-only contained) 1 drop/10 kgbw/time given 2 times a day for 12 weeks. the dose will be calculated based on body weight by the certified nutritionist during the interview after the subject signs the informed consent form
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: Propolis — intervention will use propolis extract (liquid-based) with 1 drop/10kgBW/times, 2 times in a day for 12 weeks. propolis will be given to intervention group
  Arms: Propolis
Other: placebo — intervention will use placebo with 1 drop/10kgBW/times, 2 times in a day for 12 weeks. propolis will be given control group
  Other Names: 70% caramel alcohol dye solution
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the effect of propolis administration on dysmenorrhea in endometriosis patient. the main questions it aims to answer are:

* Does the propolis administration reduce symptoms of dysmenorrhea in endometriosis?
* Does the propolis administration reduce the amount of oxidative stress biomarkers in endometriosis?
* Does the propolis administration reduce the amount of Inflammatory biomarkers in endometriosis?

Participants will be given an intervention in the form of propolis at a dose of 1 drop per 10 kilogram of body weight per administration, twice a day. there will be a control group that will be given an intervention in the form of a placebo containing 70% caramel alcohol dye solution.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 20-49 years and already menstruating with complaints of menstrual pain referred to the obstetrics and gynecology polyclinic for LNG implant placement
* Willing to have LNG implant installed after receiving explanation about implants
* Not receiving hormonal treatment for endometriosis within the last 3 months
* Can receive drops (propolis) during the study

Exclusion Criteria:

* Impaired liver function, degenerative diseases (DM, hypertension and cardiovascular disease), benign tumors, cancer
* Pregnancy and breastfeeding
* Hypersensitivity to levonogestrel
* Thromboembolic disease
* Experiencing bleeding for unknown reasons
* History of allergies to honey and its processed products
* Currently taking supplements/drugs that are not included in the standard management of endometriosis patients at RSCM
* Have consumed propolis before
* Received hormonal treatment within the last 3 months

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-06-22 (Estimated); Study Completion 2023-07-11 (Estimated)

PRIMARY OUTCOMES:
Malondialdehyde (MDA) | week 0
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using ng/mL numeric scale
Malondialdehyde (MDA) | week 4
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using ng/mL numeric scale
Malondialdehyde (MDA) | week 12
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using ng/mL numeric scale
Superoxide dismutase (SOD) | week 0
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using nmol/mLnumeric scale
Superoxide dismutase (SOD) | week 4
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using nmol/mLnumeric scale
Superoxide dismutase (SOD) | week 12
  blood biochemical test for oxidative stress biomarker from lipid peroxidation product, using nmol/mLnumeric scale
interleukin 6 | week 0
  will test the outcome with ELISA test from blood sample for inflammatory biomarker, using ng/mL numeric scale
interleukin 6 | week 4
  will test the outcome with ELISA test from blood sample for inflammatory biomarker, using ng/mL numeric scale
interleukin 6 | week 12
  will test the outcome with ELISA test from blood sample for inflammatory biomarker, using ng/mL numeric scale
tumor necrosis factor alpha (TNF alfa) | week 0
  will test the outcome with ELISA test for inflammatory biomarker, using ng/mL numeric scale
tumor necrosis factor alpha (TNF alfa) | week 4
  will test the outcome with ELISA test for inflammatory biomarker, using ng/mL numeric scale
tumor necrosis factor alpha (TNF alfa) | week 12
  will test the outcome with ELISA test for inflammatory biomarker, using ng/mL numeric scale
pain scale | week 0
  to measure the outcome, the investigators use Visual Analogue Scale for measure the pain from the subject, from 0 to 10. The scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). the subject will be asked to rate their current level of pain by placing a mark on the line.
pain scale | week 4
  to measure the outcome, the investigators use Visual Analogue Scale for measure the pain from the subject, from 0 to 10. The scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). the subject will be asked to rate their current level of pain by placing a mark on the line.
pain scale | week 12
  to measure the outcome, the investigators use Visual Analogue Scale for measure the pain from the subject, from 0 to 10. The scale consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be'). the subject will be asked to rate their current level of pain by placing a mark on the line.
Glutathione | week 0
  measure the outcome with blood biochemical test using spectrofotometri in µg/mL numeric scale
Glutathione | week 4
  measure the outcome with blood biochemical test using spectrofotometri in µg/mL numeric scale
Glutathione | week 12
  measure the outcome with blood biochemical test using spectrofotometri in µg/mL numeric scale
8-hydroxy-2-deoxyiguanosine (8-OHdG) | week 0
  measure the outcome with ELISA from blood sample in ng/mL numeric scale
8-hydroxy-2-deoxyiguanosine (8-OHdG) | week 4
  measure the outcome with ELISA from blood sample in ng/mL numeric scale
8-hydroxy-2-deoxyiguanosine (8-OHdG) | week 12
  measure the outcome with ELISA from blood sample in ng/mL numeric scale

CONTACTS AND LOCATIONS:
Overall Officials: Dwirini Retno Gunarti, Dr drg Master of Science, Principal Investigator
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta, Jakarta Pusat, Indonesia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/97/NCT05770297/Prot_ICF_001.pdf